CLINICAL TRIAL: NCT05315648
Title: The Associations Between Perioperative Depression or Anxiety, Salivary Cortisol and α-amylase, and Administered Anesthesia Type in Knee Arthroscopy With Anterior Cruciate Ligament Reconstruction (ACLR): Prospective, Randomized Trial
Brief Title: Effect of General and Non-general Anesthesia on Perioperative Depression or Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Congcong Huang, Principal Investigator, Second Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2021-03-109
Record Dates: First submitted 2021-10-26; First posted 2022-04-07 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Depression, Anxiety
Keywords: perioperative anxiety or depression; general anesthesia; salivary cortisol; salivary α-amylase; Hospital Anxiety and Depression Scale; stress response; non-general anesthesia
MeSH Terms: conditions — Depression; Anxiety Disorders; Fractures, Stress | interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio into two groups, group GA and group NGA, using a random number generator. This allocation will be written and stored in an opaque, secure envelope. Patients in group GA will receive general anesthesia followed by femoral nerve block. Patients in group NGA will receive combined spinal-epidural anesthesia followed by femoral nerve block.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both the investigator and the outcomes assessor doing follow-up interviews and extracting data from the electronic medical records will be blinded to group allocation and treatment interventions. The patients know the allocation, cause patients in group NGA will not receive any sedation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia group (Experimental): Patients in GA group will receive general anesthesia combined with FNB. All patients received routine anesthesia and surgical protocols. GA will be induced by intravenously administering propofol 2-4 mg/kg, cisatracurium 0.2mg/kg, sufentanil 0.2-0.3 μg/kg and maintained with remifentanil at 0.15-0.2 μg/kg/min and 2%-3% sevoflurane to keep bispectral index (BIS) values at 40 - 60. FNB will be performed under ultrasound-guieded and combined with nerve stimulation. Using an in-plane technique, a 10-cm long 18- gauge (G) Tuohy needle will be inserted in the lateral to medial direction towards the femoral nerve (FN). As the needle is being advanced toward the FN, the nerve stimulator is set at 1 mA, 0.1-millisecond pulse duration, and 2-Hz frequency. When the muscle contraction of the quadriceps muscle is identified, the current is reduced to 0.5 mA. After the negative aspiration, 20 mL of ropivacaine 0.375% is injected.
  Interventions: Procedure: anesthesia approach (general anesthesia or non-general anesthesia)
- Non-general anesthesia group (Experimental): Patients in NGA group will receive combined spinal-epidural anesthesia（CSEA）at L3 to L4 interspace with 3.0 ml of 0.5% hyperbaric ropivacaine followed with FNB , and without sedation. The FNB will be performed under aseptic precautions using ultrasound guidance and nerve stimulation. A high frequency linear ultrasound transducer 5-12 MHz (Sonosite, Inc. Bothell WA 98021 USA) was placed on the inguinal crease to identify the femoral artery and nerve. Using an in-plane technique, a 10-cm long 18- gauge (G) Tuohy needle connected to the nerve stimulator will be inserted in the lateral to medial direction towards the femoral nerve. When the muscle contraction of the quadriceps muscle and negative aspiration are identified, 20 mL of ropivacaine 0.375% is injected.
  If the CSEA analgesia is invalid (two times of epidural remedial analgesia) , change non-general anesthesia to general anesthesia, and the subjects withdrew from the trial.
  Interventions: Procedure: anesthesia approach (general anesthesia or non-general anesthesia)

INTERVENTIONS:
Procedure: anesthesia approach (general anesthesia or non-general anesthesia) — patients in group GA received general anesthesia followed with FNB. patients in group NGA received CSEA followed with FNB

SUMMARY:
Perioperative depression and/or anxiety play a critical role in patient presentation, satisfaction and outcomes. The aim of this study is to assess the level of perioperative depression and/or anxiety in patients with arthroscopic knee surgery and to evaluate their relationship with anesthesia approach (general anesthesia or non general anesthesia). The perioperative characteristic of depression or anxiety is assessed by Hospital Anxiety and Depression Scale (HADS) questionnaires and the level of salivary cortisol, salivary α-amylase (sAA) and blood glucose.

DETAILED DESCRIPTION:
The incidence of perioperative anxiety has been reported to range from 11% to 80% among adult patients. Perioperative depression and/or anxiety may increase the risk of poor postoperative outcomes including increased morbidity and mortality , increased health care utilization, increased opioid consumptions and pain scores, and decreased quality of recovery. Previous studies have found that worrying about postoperative pain, unease of separation from family, loss of selfcare and work ability, fear of surgery and even death are common factors leading to perioperative anxiety symptoms.

The investigators found there were not enough studies to gain insights into the public's knowledges, attitudes, and concerns regarding the risks associated with anesthesia. To some, the fear of general anesthesia (GA) remains prevalent, especially with regard to possible brain damage, death, and intraoperative awareness. The others, neuraxial anesthesia was supposed to result in potentially complications, including postdural puncture headache, backache, transient neurological symptoms, epidural hematoma and abscess, meningitis, arachnoiditis, postoperative urinary retention, local anesthetic systemic toxicity.

Such fears can even exceed the anxiety about actual surgery. Actually, anesthesia approach can be selected based on patients and anesthesiologists preference.

The investigators assumed from clinical experiences that effects of different anesthetic approach and anesthetic drugs on stress reaction, perioperative blood glucose, immunity or neuroendocrine during surgical operation were different, which resulted different prognosis of patients.

The perioperative characteristic of depression or anxiety is assessed by Hospital Anxiety and Depression Scale (HADS) questionnaires, salivary cortisol, salivary α-amylase (sAA) and blood glucose.

Salivary cortisol and a-amylase are produced respectively by the hypothalamus-pituitary-adrenal (HPA) axis and the sympathetic-adrenomedullary (SAM) system during stress response, still not included in the routine evaluation of perioperative physiological stress response. The application of these tests require additional and definitive validation. In our study, salivary cortisol and a-amylase are measured as stress biomarkers to examine their associations with anesthetic approach.The correlation between salivary cortisol and serum cortisol was excellent in dynamic tests of adrenal function (dexamethasone suppression, adreno-cortico-tropic-hormone stimulation), in healthy subjects and in patients with adrenal insufficiency, in tests of circadian variation and in randomly collected samples. The rate of equilibrium of cortisol between blood and saliva was very fast, being less than 5 minutes. Since only free levels of cortisol are detected in saliva, salivary cortisol is suggested to be a more appropriate measure for the clinical assessment of adrenocortical function than serum cortisol. sAA has been proposed as a sensitive biomarker for stress-related changes in the body that reflect the activity of the sympathetic nervous system, and a growing body of research is accumulating to support the validity and reliability of this parameter. Numerous studies applying stress protocols have demonstrated that salivary a-amylase is highly sensitive to stress-related changes.

The investigators are trying to recruit patients who are scheduled to undergo knee arthroscopy with anterior cruciate ligament reconstruction (ACLR) for the first time. Those patients will be randomly assigned to general anesthesia (GA) group or non-general anesthesia (NGA) group. Patients in GA group will received general anesthesia combined with femoral nerve block (FNB). Patients in NGA group will received neuraxial anesthesia combined with FNB, and without sedation. All patients received routine anesthesia and surgical protocols and will be sent to the postoperative recovery unit (PACU) after surgery. Intraoperative vital signs, analgesic usage, and duration of surgery were recorded.

The primary outcomes are HADS scores , salivary cortisol, sAA, blood glucose，swelling ratings postoperatively, temperature ratings postoperatively and hospital stay. Secondary outcomes are analgesic usage intraoperative and postoperative, anesthesia induction pain score, postoperative pain score, duration of stay in the recovery unit, incidences of complications about relevant anesthesia.

The Patients Hospital Anxiety and Depression Scale (HADS), a 14-item scale (7 items each for anxiety and depression), with each item scored from 0 to 3. Salivary cortisol, sAA and blood glucose levels will be tested in the morning one day before operation (T0), on the day of operation (T1), 2 hours after operation (T2), the first morning after operation (T3), the second morning after operation (T4).

The investigators will conduct subgroup analysis based on the patients' anesthesia wishes (conform to patient's wishes, against patient's wishes, no original opinion) to address the influence of anaesthesia practice and perioperative stress response.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be scheduled to receive anterior cruciate ligament reconstruction of knee joint for the first time
* American Society of Anesthesiologists (ASA) physical status I or II
* The operation time is less than 2 hours (from the beginning use of the tourniquet to the release)

Exclusion Criteria:

* Clinical diagnosis of anxiety or depression or mania
* Clinical diagnosis of systemic diseases (systemic sclerosis, systemic lupus erythematosus, rheumatoid arthritis, rheumatoid arthritis, primary aldosteronism, Cushing syndrome)
* Medication history of cortisol or sedative hypnotic drugs
* Tumor patients
* Smoking
* Pregnancy status
* Diabetes
* Drinking coffee or alcohol drinks during perioperative period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
The rate of Anxiety symptoms (HADS-A) | one day before surgery, 1day, 3 days after surgery and 5 days after surgery while in hospital
  The HADS scale includes two dimensions of anxiety and depression, with a total of 14 items, 7 items for anxiety and 7 items for depression.
  The score for each individual item could vary from 0 to 3, so that the total score for each scale about anxiety (HADS-A) ranges from 0 to 21. If the score was 0-7, indicating that there was no anxiety; the score was 8-10, suspected anxiety; 11-14, moderate anxiety; the score was 15-21, severe anxiety. If the score is ≥ 8, it will be rated as positive, otherwise it will be rated as negative.
The rate of Depression symptoms (HADS-D) | one day before surgery, 1day, 3 days after surgery and 5 days after surgery while in hospital
  The HADS scale includes two dimensions of anxiety and depression, with a total of 14 items, 7 items for anxiety and 7 items for depression.
  The score for each individual item could vary from 0 to 3, so that the total score for each scale about depression (HADS-D) ranges from 0 to 21. If the score was 0-7, indicating that there was no depression; the score was 8-10, suspected depression; 11-14, moderate depression; the score was 15-21, severe depression. If the score is ≥ 8, it will be rated as positive, otherwise it will be rated as negative.
The changes of salivary cortisol concentration | on the day of surgery (6 - 8 am), at 2 hours after surgery, the first morning after surgery (6 - 8 am) and the second morning after surgery (6 - 8 am)
  Enzyme immunoassay for the quantitative determination of free Cortisol in human saliva.The patient should not eat, drink, chew gums or brush teeth for 30 min before sampling.Otherwise rinse mouth thoroughly with cold water 5 min prior to sample collection.A minimum of 0.5 mL liquid should be collected. Saliva flow can be stimulated by chewing on a piece of Parafilm.
The changes of Saliva α- amylase activity | on the day of surgery (6 - 8 am), at 2 hours after surgery, the first morning after surgery (6 - 8 am) and the second morning after surgery (6 - 8 am)
  Enzymatic assay for the determination of alpha amylase activity in human saliva.The patient should not eat, drink, chew gums or brush teeth for 30 min before sampling.Otherwise rinse mouth thoroughly with cold water 5 min prior to sample collection.A minimum of 0.5 mL liquid should be collected. Saliva flow can be stimulated by chewing on a piece of Parafilm.
The changes of Blood glucose level | on the day of surgery (6 - 8 am), at 2 hours after surgery, the first morning after surgery (6 - 8 am) and the second morning after surgery (6 - 8 am)
  Using a glucose meter to check and monitor blood sugar via finger stick

SECONDARY OUTCOMES:
The changes of swelling rating | at 6, 12, 24, 48, and 72 hours after surgery
  The postoperative knee swelling rating on the surgical side is defined as the knee circumference on the surgical side minus the knee circumference on the non-suigical side, both measured in centimeters (cm) at 5.08 cm above the superior border of the patella, 6 h, 12 h, 24 h, 48 h, and 72 h postoperatively. The larger value means more severe swelling after surgery.
Post-operative opioid consumptions | from arrived at PACU to the first 72 post-operative hours
  postoperative opioid consumption including sufentanil consumptions in PACU and the rescue analgesics (morphine 0.05 mg/kg) when NRS > 3. (sufentanil will be converted into morphine equivalents)
The changes of NRS of postoperative pain | at 2, 6, 12, 24, 48, and 72 hours after surgery
  Patients evaluate the pain at rest and on knee flexion after surgery. NRS will be used to assess the intensity of pain, ranged from 0-10, 0 means no pain and 10 means severe pain.
Complications related to general anesthesia | started from the induction of general anesthesia to the first 72 post-operative hours
  Number of Participants with the complications relaterd to general anesthesia such as intraoperative hypoxemia, postoperative nausea and vomiting , postoperative deliriums, postoperative cognitive dysfunction in each group
Complications related to combined spinal-epidural anesthesia | started from the beginning of combined spinal-epidural anesthesia to the first 72 post-operative hours
  Number of Participants with the complications relaterd to combined spinal-epidural anesthesia such as postdural puncture headache, backache, transient neurological symptoms, epidural hematoma and abscess, meningitis, arachnoiditis, postoperative urinary retention, local anesthetic systemic toxicity and infection in each group
Complications related to femoral nerve block | started from the puncture of nerve block to the first 72 post-operative hours
  Number of Participants with the complications relaterd to femoral nerve block such as nerve injury, hematoma, local anesthetic systemic toxicity and infection in each group
Costs of hospitalization | through study completion, an average of 1 week
  Costs will be calculated about total standardized costs before healthcare coverage，such as social medical reimbursement or health insurance.Costs will be evaluated in 2022 renminbi (RMB) yuans.
The changes of skin temperature rating | at 1, 3, and 5 days after surgery
  Skin temperature of the knee is measured at the center of the anterior patella on postoperative days 1, 3, and 5. Limbs will be exposed to room temperature for 5 minutes bilaterally and then the skin temperature was measured with a skin temperature gun. The skin temperature on the surgical side was defined as the skin temperature on the surgical side minus the skin temperature on the unsurgical side, both measured in degrees centigrade (°C) .
Length of hospital stay | The length of hospital stay was counted in days, about 5 to 7 days usually
  from the day when the patients arrived at the ward for reception to the day when the patients discharged, based on the electronic medical record system

CONTACTS AND LOCATIONS:
Overall Officials: CongCong Huang, Master, Study Director — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- Second Affiliated Hospital of WenZhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khoo B, Boshier PR, Freethy A, Tharakan G, Saeed S, Hill N, Williams EL, Moorthy K, Tolley N, Jiao LR, Spalding D, Palazzo F, Meeran K, Tan T. Redefining the stress cortisol response to surgery. Clin Endocrinol (Oxf). 2017 Nov;87(5):451-458. doi: 10.1111/cen.13439. Epub 2017 Aug 30. PMID 28758231
- [Background] Nagase K, Ando-Nagase K. Preoperative anxiety and intraoperative anesthetic requirements. Anesth Analg. 2000 Jul;91(1):250. doi: 10.1097/00000539-200007000-00062. No abstract available. PMID 10866931
- [Background] Takagi H, Ando T, Umemoto T; ALICE (All-Literature Investigation of Cardiovascular Evidence) Group. Perioperative depression or anxiety and postoperative mortality in cardiac surgery: a systematic review and meta-analysis. Heart Vessels. 2017 Dec;32(12):1458-1468. doi: 10.1007/s00380-017-1022-3. Epub 2017 Jul 13. PMID 28702898
- [Background] Dunn LK, Durieux ME, Fernandez LG, Tsang S, Smith-Straesser EE, Jhaveri HF, Spanos SP, Thames MR, Spencer CD, Lloyd A, Stuart R, Ye F, Bray JP, Nemergut EC, Naik BI. Influence of catastrophizing, anxiety, and depression on in-hospital opioid consumption, pain, and quality of recovery after adult spine surgery. J Neurosurg Spine. 2018 Jan;28(1):119-126. doi: 10.3171/2017.5.SPINE1734. Epub 2017 Nov 10. PMID 29125426
- [Background] Smith PJ, Snyder LD, Palmer SM, Hoffman BM, Stonerock GL, Ingle KK, Saulino CK, Blumenthal JA. Depression, social support, and clinical outcomes following lung transplantation: a single-center cohort study. Transpl Int. 2018 May;31(5):495-502. doi: 10.1111/tri.13094. Epub 2017 Dec 14. PMID 29130541
- [Background] Caumo W, Schmidt AP, Schneider CN, Bergmann J, Iwamoto CW, Bandeira D, Ferreira MB. Risk factors for preoperative anxiety in adults. Acta Anaesthesiol Scand. 2001 Mar;45(3):298-307. doi: 10.1034/j.1399-6576.2001.045003298.x. PMID 11207465
- [Background] Capdevila X, Dadure C. Perioperative management for one day hospital admission: regional anesthesia is better than general anesthesia. Acta Anaesthesiol Belg. 2004;55 Suppl:33-6. PMID 15625956
- [Background] Johnson RL, Kopp SL, Burkle CM, Duncan CM, Jacob AK, Erwin PJ, Murad MH, Mantilla CB. Neuraxial vs general anaesthesia for total hip and total knee arthroplasty: a systematic review of comparative-effectiveness research. Br J Anaesth. 2016 Feb;116(2):163-76. doi: 10.1093/bja/aev455. PMID 26787787
- [Background] Imbelloni LE, Fornasari M, Fialho JC, Sant'Anna R, Cordeiro JA. General anesthesia versus spinal anesthesia for laparoscopic cholecystectomy. Rev Bras Anestesiol. 2010 May-Jun;60(3):217-27. doi: 10.1016/S0034-7094(10)70030-1. PMID 20682154
- [Background] Wu L, Zhao H, Wang T, Pac-Soo C, Ma D. Cellular signaling pathways and molecular mechanisms involving inhalational anesthetics-induced organoprotection. J Anesth. 2014 Oct;28(5):740-58. doi: 10.1007/s00540-014-1805-y. Epub 2014 Mar 9. PMID 24610035
- [Background] Edipoglu IS, Celik F. The Associations Between Cognitive Dysfunction, Stress Biomarkers, and Administered Anesthesia Type in Total Knee Arthroplasties: Prospective, Randomized Trial. Pain Physician. 2019 Sep;22(5):495-507. PMID 31561651
- [Background] Franks NP. Molecular targets underlying general anaesthesia. Br J Pharmacol. 2006 Jan;147 Suppl 1(Suppl 1):S72-81. doi: 10.1038/sj.bjp.0706441. PMID 16402123
- [Background] Chau PL. New insights into the molecular mechanisms of general anaesthetics. Br J Pharmacol. 2010 Sep;161(2):288-307. doi: 10.1111/j.1476-5381.2010.00891.x. PMID 20735416
- [Background] Cozma S, Dima-Cozma LC, Ghiciuc CM, Pasquali V, Saponaro A, Patacchioli FR. Salivary cortisol and alpha-amylase: subclinical indicators of stress as cardiometabolic risk. Braz J Med Biol Res. 2017 Feb 6;50(2):e5577. doi: 10.1590/1414-431X20165577. PMID 28177057
- [Background] Burke HM, Davis MC, Otte C, Mohr DC. Depression and cortisol responses to psychological stress: a meta-analysis. Psychoneuroendocrinology. 2005 Oct;30(9):846-56. doi: 10.1016/j.psyneuen.2005.02.010. PMID 15961250
- [Background] Hellhammer DH, Wust S, Kudielka BM. Salivary cortisol as a biomarker in stress research. Psychoneuroendocrinology. 2009 Feb;34(2):163-171. doi: 10.1016/j.psyneuen.2008.10.026. Epub 2008 Dec 18. PMID 19095358
- [Background] Jezova D, Trebaticka J, Buzgoova K, Durackova Z, Hlavacova N. Lower activity of salivary alpha-amylase in youths with depression. Stress. 2020 Nov;23(6):688-693. doi: 10.1080/10253890.2020.1777975. Epub 2020 Jun 22. PMID 32510266
- [Background] Benson S, Siebert C, Koenen LR, Engler H, Kleine-Borgmann J, Bingel U, Icenhour A, Elsenbruch S. Cortisol affects pain sensitivity and pain-related emotional learning in experimental visceral but not somatic pain: a randomized controlled study in healthy men and women. Pain. 2019 Aug;160(8):1719-1728. doi: 10.1097/j.pain.0000000000001579. PMID 31335642
- [Background] Ezhevskaya AA, Mlyavykh SG, Anderson DG. Effects of continuous epidural anesthesia and postoperative epidural analgesia on pain management and stress response in patients undergoing major spinal surgery. Spine (Phila Pa 1976). 2013 Jul 1;38(15):1324-30. doi: 10.1097/BRS.0b013e318290ff26. PMID 23514874
- [Background] Wang J, Yin Y, Zhu Y, Xu P, Sun Z, Miao C, Zhong J. Thoracic epidural anaesthesia and analgesia ameliorates surgery-induced stress response and postoperative pain in patients undergoing radical oesophagectomy. J Int Med Res. 2019 Dec;47(12):6160-6170. doi: 10.1177/0300060519866943. Epub 2019 Aug 19. PMID 31426685
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Delle Chiaie R, Trabucchi G, Girardi N, Marini I, Pannese R, Vergnani L, Caredda M, Zerella MP, Minichino A, Corrado A, Patacchioli FR, Simeoni S, Biondi M. Group psychoeducation normalizes cortisol awakening response in stabilized bipolar patients under pharmacological maintenance treatment. Psychother Psychosom. 2013;82(4):264-6. doi: 10.1159/000348609. Epub 2013 Jun 1. No abstract available. PMID 23736884
- [Background] Ghiciuc CM, Dima Cozma LC, Bercea RM, Lupusoru CE, Mihaescu T, Szalontay A, Gianfreda A, Patacchioli FR. Restoring the salivary cortisol awakening response through nasal continuous positive airway pressure therapy in obstructive sleep apnea. Chronobiol Int. 2013 Oct;30(8):1024-31. doi: 10.3109/07420528.2013.795155. Epub 2013 Jul 16. PMID 23859257
- [Background] Schumacher S, Kirschbaum C, Fydrich T, Strohle A. Is salivary alpha-amylase an indicator of autonomic nervous system dysregulations in mental disorders?--a review of preliminary findings and the interactions with cortisol. Psychoneuroendocrinology. 2013 Jun;38(6):729-43. doi: 10.1016/j.psyneuen.2013.02.003. Epub 2013 Mar 5. PMID 23481259
- [Background] Blair J, Adaway J, Keevil B, Ross R. Salivary cortisol and cortisone in the clinical setting. Curr Opin Endocrinol Diabetes Obes. 2017 Jun;24(3):161-168. doi: 10.1097/MED.0000000000000328. PMID 28375882
- [Background] Proctor GB, Carpenter GH. Regulation of salivary gland function by autonomic nerves. Auton Neurosci. 2007 Apr 30;133(1):3-18. doi: 10.1016/j.autneu.2006.10.006. Epub 2006 Dec 6. PMID 17157080
- [Background] DeCaro JA. Methodological considerations in the use of salivary alpha-amylase as a stress marker in field research. Am J Hum Biol. 2008 Sep-Oct;20(5):617-9. doi: 10.1002/ajhb.20795. PMID 18491409
- [Background] Thapa D, Ahuja V, Verma P, Gombar S, Gupta R, Dhiman D. Post-operative analgesia using intermittent vs. continuous adductor canal block technique: a randomized controlled trial. Acta Anaesthesiol Scand. 2016 Nov;60(10):1379-1385. doi: 10.1111/aas.12787. Epub 2016 Sep 4. PMID 27592690
- [Background] Abdallah FW, Mejia J, Prasad GA, Moga R, Chahal J, Theodoropulos J, Dwyer T, Brull R. Opioid- and Motor-sparing with Proximal, Mid-, and Distal Locations for Adductor Canal Block in Anterior Cruciate Ligament Reconstruction: A Randomized Clinical Trial. Anesthesiology. 2019 Sep;131(3):619-629. doi: 10.1097/ALN.0000000000002817. PMID 31246607
- [Background] Ogura T, Omatsu H, Fukuda H, Asai S, Saito C, Takahashi T, Ichino Y, Omodani T, Sakai H, Yamaura I, Kawasaki Y, Tsuchiya A, Takahashi K. Femoral nerve versus adductor canal block for early postoperative pain control and knee function after anterior cruciate ligament reconstruction with hamstring autografts: a prospective single-blind randomised controlled trial. Arch Orthop Trauma Surg. 2021 Nov;141(11):1927-1934. doi: 10.1007/s00402-021-03823-1. Epub 2021 Feb 20. PMID 33609182
- [Background] Louise Fincher A, William Woods G, O'Connor DP. Intraoperative Arthroscopic Cold Irrigation Solution Does Not Affect Postoperative Pain and Swelling. J Athl Train. 2004 Mar;39(1):12-16. PMID 15085206